CLINICAL TRIAL: NCT01621165
Title: Prazosin as an Antimanic Agent in Severe Mania or Mixed Episodes: a Double-blind, Placebo-controlled Study
Brief Title: Prazosin as an Antimanic Agent in Severe Mania or Mixed States
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to recruit subjects given short length of stay in hospital
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Elizabeth S. Liebson, PI, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12909
Record Dates: First submitted 2009-03-17; First posted 2012-06-18 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2012-06

CONDITIONS: Bipolar, Mania; Bipolar, Mixed State
Keywords: treatment of bipolar, mania; double-blind, placebo-controlled study; drug intervention; add-on study; prazosin; alpha-1 adrenergic antagonist
MeSH Terms: conditions — Mania | interventions — Prazosin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- prazosin (Active Comparator): Add prazosin to usual medications and monitor manic symptoms and for adverse effects
  Interventions: Drug: Addition of prazosin to usual care (add-on study)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Addition of prazosin to usual care (add-on study) — Prazosin and placebo will be gradually titrated over 10 days to a final dose of 10 mg/day, given in divided doses (three times a day). During this time subjects will be monitored for adverse effects to prazosin and manic symptoms will be monitored. Vital signs will be monitored three times a day throughout the study. If a subject receiving prazosin or placebo develops distressing adverse effects, the dose will be decreased to the next lower dose.If there is a greater than 15 mg mercury postural fall in systolic bBP, dosing will be held at the previous day's dose.Subjects who do not tolerate prazosin or placebo will be discharged from the study.
  Other Names: Minipress
  Arms: prazosin
Drug: Placebo — Prazosin and placebo will be gradually titrated over 10 days to a final dose of 10 mg/day, given in divided doses (three times a day). During this time subjects will be monitored for adverse effects to prazosin and manic symptoms will be monitored. Vital signs will be monitored three times a day throughout the study. If a subject receiving prazosin or placebo develops distressing adverse effects, the dose will be decreased to the next lower dose.If there is a greater than 15 mg mercury postural fall in systolic bBP, dosing will be held at the previous day's dose.Subjects who do not tolerate prazosin or placebo will be discharged from the study.
  Arms: Placebo

SUMMARY:
Mania has been considered to be, in part, a hyperadrenergic state. One focus of treatment of mania involves directly targeting this hyperexcitable state by reducing arousal with antiadrenergic agents. This can be achieved by decreasing norepinephrine release by stimulating presynaptic inhibitory receptors. Prazosin, FDA approved for the treatment of high blood pressure works in part by blocking postsynaptic alpha-adrenergic receptors. Prazosin has been found to be clinically useful for the treatment of Post Traumatic Stress Disorder. It is reasonable, therefore, to anticipate that prazosin might be helpful in the treatment of mania.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60
* Primary diagnosis of bipolar disorder with severe mania or mixed episode
* YMRS score of > 20
* Documented medical evaluation without acute or serious medical illness
* Negative pregnancy test
* Healthy functioning liver

Exclusion Criteria:

* Lack of capacity to provide informed consent
* Involuntary commitment
* Low blood pressure
* History of adverse reaction or allergy to prazosin or other quinazolines
* Informed consent not given or retracted during study
* History of narcolepsy
* Unstable or acute medical illness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Young Mania Rating Scale (YMRS) | 10 days

SECONDARY OUTCOMES:
Mania Acute Changes Scale (MACS) | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth S Liebson, MD, Principal Investigator — Mclean Hospital